CLINICAL TRIAL: NCT01634152
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group Trial to Evaluate Efficacy and Safety of Tiotropium Inhalation Solution (2.5 mcg and 5 mcg) Delivered Via Respimat® Inhaler Once Daily in the Evening Over 12 Weeks as add-on Controller Therapy on Top of Usual Care in Children (6 to 11 Years Old) With Severe Persistent Asthma
Brief Title: Efficacy and Safety of 2 Doses of Tiotropium Respimat® Compared to Placebo in Children With Severe Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.446; 2011-001777-43 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

ARMS (3):
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo
- Tiotropium low dose QD (Experimental)
  Interventions: Drug: Tiotropium low dose mcg
- Tiotropium medium dose QD (Experimental)
  Interventions: Drug: Tiotropium high dose

INTERVENTIONS:
Drug: Placebo — 2 actuations once daily in the evening
  Arms: Placebo QD
Drug: Tiotropium low dose mcg — 2 actuations once daily in the evening
  Arms: Tiotropium low dose QD
Drug: Tiotropium high dose — 2 actuations once daily in the evening
  Arms: Tiotropium medium dose QD

SUMMARY:
The overall purpose of the trial is to evaluate efficacy and safety of tiotropium inhalation solution (2.5 mcg and 5 mcg) delivered via Respimat® inhaler once daily in the evening over 12 weeks, compared to placebo, as add-on controller therapy on top of usual care in children (6 to 11 years old) with severe persistent asthma.

ELIGIBILITY:
Inclusion criteria:

Inclusion criteria are:

1. All patients' parent(s) (or legal guardian) must sign and date an informed consent prior to participation in the trial. In addition, an informed assent suitable for this age group has to be obtained from patients. A separate informed consent/assent is required for pharmacogenomic sampling.
2. Male or female patients between 6 and 11 years of age.
3. All patients must have at least a 6-month history of asthma.
4. All patients must have been on maintenance treatment with an inhaled corticosteroid either at stable high dose in combination with another controller medication, OR at stable medium dose in combination with two other controller medications, for at least 4 weeks before Visit 1.
5. All patients must be symptomatic (partly controlled) at Visit 1 and prior to randomisation at Visit 2 as defined by an Asthma Control Questionnaire (ACQ-IA) mean score >= 1.5.
6. All patients must have a pre-bronchodilator forced expiratory volume in one second (FEV1) >= 60% and <= 90% of predicted normal at Visit 1.
7. Variation of absolute FEV1 values of Visit 1 (pre-bronchodilator, considered as 100%) as compared to Visit 2 (pre-dose) must be within ± 30%.
8. All patients must confirm the diagnosis of asthma by bronchodilator reversibility at Visit 1, resulting in an increase in FEV1 of >= 12% 15 to 30 minutes after 200 mcg salbutamol/albuterol.
9. Patients must be able to use the Respimat inhaler correctly.
10. Patients must be able to perform all trial related procedures including technically acceptable pulmonary function tests and use of electronic diary/peak flow meter (diary compliance of at least 80% is required).

Exclusion criteria:

Exclusion criteria are:

1. Patients with a significant disease other than asthma.
2. Patients with a clinically relevant abnormal haematology or blood chemistry at screening.
3. Patients with a history of congenital or acquired heart disease, or patients who have been hospitalised for cardiac syncope or failure during the past year.
4. Patients with any unstable or life-threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year.
5. Patients with a malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years.
6. Patients with known active tuberculosis.
7. Patients who have undergone thoracotomy with pulmonary resection.
8. Patients who are currently in a pulmonary rehabilitation program or have completed a pulmonary rehabilitation program in the six weeks prior to Visit 1.
9. Patients with known hypersensitivity to anticholinergic drugs, BAC, EDTA or any other components of the inhalation solution used with the Respimat inhaler.
10. Pregnant or nursing female patients, including postmenarchal girls with a positive urine pregnancy test at Visit 1.
11. Postmenarchal girls of child-bearing potential not using a highly effective method of birth control.
12. Patients who have been treated with systemic corticosteroids within four weeks prior to Visit 1.
13. Patients who have been treated with systemic beta-adrenergics within four weeks prior to Visit 1.
14. Patients who have been treated with oral beta-blocker medication within four weeks prior to Visit 1 and/or during the screening period.
15. Patients who have been treated with inhaled long-acting anticholinergics or systemic anticholinergic treatment within four weeks prior to Visit 1 and/or during the screening period, or who have been treated with inhaled short-acting anticholinergics within two weeks prior to Visit 1.
16. Patients who have been treated with short-acting theophylline preparations within two weeks prior to Visit 1.
17. Patients who have been treated with non-approved and according to international guidelines not recommended experimental drugs for routine asthma therapy within four weeks prior to Visit 1 and/or during the screening period.
18. Patients who have taken an investigational drug within six half lives according to the investigator's information, or four weeks (whichever is greater) prior to Visit 1 and/or during the screening period.
19. Patients who have previously been randomised in this trial or are currently participating in another trial.
20. Patients with any acute asthma exacerbation or respiratory tract infection in the four weeks prior to Visit 1 and/or in the four weeks prior to Visit 2. In case of an asthma deterioration occurring in the four weeks prior to Visit 1 and/or in the four weeks prior to Visit 2, the visit must be postponed.
21. Patients requiring six or more puffs of rescue medication per day on more than two consecutive days in the four weeks prior to Visit 1 and/or in the four weeks prior to Visit 2. In case of an asthma deterioration occurring in the four weeks prior to Visit 1 and/or in the four weeks prior to Visit 2, the visit must be postponed.
22. Patients who are unable to comply with medication restrictions prior to Visit 1 and/or prior to Visit 2.
23. Patients with a known narrow-angle glaucoma, or any other disease where anticholinergic treatment is contraindicated.
24. Patients with moderate to severe renal impairment, as defined by a creatinine clearance <50 mL/min/1.73 m2 BSA, as tiotropium is a predominantly renally excreted drug.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 401 (Actual)
Dates: Start 2012-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (94):
- United States (10):
  - 205.446.01014 Boehringer Ingelheim Investigational Site, Rolling Hills Estates, California
  - 205.446.01011 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 205.446.01003 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 205.446.01009 Boehringer Ingelheim Investigational Site, Columbia, Missouri
  - 205.446.01005 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.446.01010 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 205.446.01004 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 205.446.01002 Boehringer Ingelheim Investigational Site, North Charleston, South Carolina
  - 205.446.01012 Boehringer Ingelheim Investigational Site, Arlington, Texas
  - 205.446.01013 Boehringer Ingelheim Investigational Site, San Antonio, Texas
- Argentina (7):
  - 205.446.54006 Boehringer Ingelheim Investigational Site, Buenos Aires
  - 205.446.54002 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.446.54003 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.446.54008 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.446.54005 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 205.446.54004 Boehringer Ingelheim Investigational Site, Mendoza
  - 205.446.54007 Boehringer Ingelheim Investigational Site, San Miguel de Tucumán
- Australia (2):
  - 205.446.61003 Boehringer Ingelheim Investigational Site, Herston, Queensland
  - 205.446.61001 Boehringer Ingelheim Investigational Site, Perth, Western Australia
- Belgium (3):
  - 205.446.32004 Boehringer Ingelheim Investigational Site, Antwerp
  - 205.446.32005 Boehringer Ingelheim Investigational Site, Bruges
  - 205.446.32006 Boehringer Ingelheim Investigational Site, Namur
- Brazil (7):
  - 205.446.55001 Boehringer Ingelheim Investigational Site, Curitiba
  - 205.446.55007 Boehringer Ingelheim Investigational Site, Goiânia
  - 205.446.55006 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 205.446.55002 Boehringer Ingelheim Investigational Site, São Paulo
  - 205.446.55003 Boehringer Ingelheim Investigational Site, São Paulo
  - 205.446.55004 Boehringer Ingelheim Investigational Site, São Paulo
  - 205.446.55005 Boehringer Ingelheim Investigational Site, São Paulo
- Canada (2):
  - 205.446.02003 Boehringer Ingelheim Investigational Site, London, Ontario
  - 205.446.02001 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
- Czechia (4):
  - 205.446.42005 Boehringer Ingelheim Investigational Site, Jablonec nad Nisou
  - 205.446.42001 Boehringer Ingelheim Investigational Site, Jihlava
  - 205.446.42002 Boehringer Ingelheim Investigational Site, Prague
  - 205.446.42004 Boehringer Ingelheim Investigational Site, Prague
- Germany (8):
  - 205.446.49012 Boehringer Ingelheim Investigational Site, Berlin
  - 205.446.49015 Boehringer Ingelheim Investigational Site, Berlin
  - 205.446.49001 Boehringer Ingelheim Investigational Site, Bochum
  - 205.446.49007 Boehringer Ingelheim Investigational Site, Dresden
  - 205.446.49003 Boehringer Ingelheim Investigational Site, Frankfurt
  - 205.446.49009 Boehringer Ingelheim Investigational Site, Koblenz
  - 205.446.49014 Boehringer Ingelheim Investigational Site, Marburg
  - 205.446.49011 Boehringer Ingelheim Investigational Site, Mönchengladbach
- Guatemala (4):
  - 205.446.50201 Boehringer Ingelheim Investigational Site, Guatemala City
  - 205.446.50202 Boehringer Ingelheim Investigational Site, Guatemala City
  - 205.446.50203 Boehringer Ingelheim Investigational Site, Guatemala City
  - 205.446.50204 Boehringer Ingelheim Investigational Site, Guatemala City
- Hungary (4):
  - 205.446.36002 Boehringer Ingelheim Investigational Site, Ajka
  - 205.446.36001 Boehringer Ingelheim Investigational Site, Budapest
  - 205.446.36003 Boehringer Ingelheim Investigational Site, Nagyatád
  - 205.446.36004 Boehringer Ingelheim Investigational Site, Szeged
- Latvia (8):
  - 205.446.37105 Boehringer Ingelheim Investigational Site, Baldone
  - 205.446.37104 Boehringer Ingelheim Investigational Site, Balvi
  - 205.446.37108 Boehringer Ingelheim Investigational Site, Daugavpils
  - 205.446.37107 Boehringer Ingelheim Investigational Site, Jēkabpils
  - 205.446.37101 Boehringer Ingelheim Investigational Site, Ogre
  - 205.446.37106 Boehringer Ingelheim Investigational Site, Rēzekne
  - 205.446.37102 Boehringer Ingelheim Investigational Site, Riga
  - 205.446.37103 Boehringer Ingelheim Investigational Site, Riga
- Lithuania (4):
  - 205.446.37004 Boehringer Ingelheim Investigational Site, Šiauliai
  - 205.446.37003 Boehringer Ingelheim Investigational Site, Tauragė
  - 205.446.37002 Boehringer Ingelheim Investigational Site, Utena
  - 205.446.37001 Boehringer Ingelheim Investigational Site, Vilnius
- Poland (4):
  - 205.446.48004 Boehringer Ingelheim Investigational Site, Bialystok
  - 205.446.48002 Boehringer Ingelheim Investigational Site, Lodz
  - 205.446.48001 Boehringer Ingelheim Investigational Site, Lublin
  - 205.446.48003 Boehringer Ingelheim Investigational Site, Tarnów
- 205.446.40002 Boehringer Ingelheim Investigational Site, Bucharest, Romania
- Russia (10):
  - 205.446.70002 Boehringer Ingelheim Investigational Site, Moscow
  - 205.446.70005 Boehringer Ingelheim Investigational Site, Moscow
  - 205.446.70007 Boehringer Ingelheim Investigational Site, Moscow
  - 205.446.70011 Boehringer Ingelheim Investigational Site, Moscow
  - 205.446.70012 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 205.446.70001 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.446.70003 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.446.70004 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.446.70010 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.446.70009 Boehringer Ingelheim Investigational Site, Yaroslavl
- Slovakia (3):
  - 205.446.42101 Boehringer Ingelheim Investigational Site, Košice
  - 205.446.42103 Boehringer Ingelheim Investigational Site, Prešov
  - 205.446.42102 Boehringer Ingelheim Investigational Site, Spišská Nová Ves
- Ukraine (13):
  - 205.446.38013 Boehringer Ingelheim Investigational Site, Chernivtsi
  - 205.446.38002 Boehringer Ingelheim Investigational Site, Dnipropetrovsk
  - 205.446.38003 Boehringer Ingelheim Investigational Site, Dnipropetrovsk
  - 205.446.38005 Boehringer Ingelheim Investigational Site, Donetsk
  - 205.446.38012 Boehringer Ingelheim Investigational Site, Donetsk
  - 205.446.38009 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.446.38004 Boehringer Ingelheim Investigational Site, Kiev
  - 205.446.38006 Boehringer Ingelheim Investigational Site, Kryvyi Rih
  - 205.446.38001 Boehringer Ingelheim Investigational Site, Lviv
  - 205.446.38014 Boehringer Ingelheim Investigational Site, Odesa
  - 205.446.38010 Boehringer Ingelheim Investigational Site, Vinnytsia
  - 205.446.38011 Boehringer Ingelheim Investigational Site, Zaporizhya
  - 205.446.38008 Boehringer Ingelheim Investigational Site, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Respimat: Inhalation of placebo solution (2 puffs) once daily for 12 weeks delivered by the Respimat inhaler, as add on therapy on top of usual care.
- Tio R2.5: Inhalation of 2.5mcg tiotropium (Tio R2.5) solution (2 puffs of 1.25mcg) once daily for 12 weeks delivered by the Respimat inhaler, as add on therapy on top of usual care.
- Tio R5: Inhalation of 5mcg tiotropium (Tio R5) solution (2 puffs of 2.5mcg) once daily for 12 weeks delivered by the Respimat inhaler, as add on therapy on top of usual care.
Period: Overall Study
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Started | 134 | 137 | 130
Completed | 130 | 136 | 126
Not Completed | 4 | 1 | 4
Not completed — Adverse Event | 2 | 0 | 2
Not completed — Consent withdrawn not due to AE | 1 | 0 | 1
Not completed — Not treated | 0 | 1 | 0
Not completed — Other reason not defined above | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set which included all randomised patients who were dispensed study medication and were documented to have taken at least 1 dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5 | Total
Number analyzed (Participants) | 134 | 136 | 130 | 400
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.1 (1.6) | 8.8 (1.7) | 9.2 (1.6) | 9.0 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 40 | 40 | 121
  Male | 93 | 96 | 90 | 279

OUTCOME MEASURES:

1. Primary Outcome: FEV1 Peak(0-3h) Change From Baseline
Description: Change from baseline in peak forced expiratory volume in 1 second within the first 3 hours post dosing (FEV1 peak(0-3h)) measured at week 12.
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: Full Analysis Set (FAS) was the same as the treated set which included all randomised patients who were dispensed and received at least one documented dose of trial medication. Missing data at a visit was imputed by the available data from the patient at that visit. Completely missing data were handled by the statistical model.
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 130 | 135 | 128
Litres | 0.252 (0.025) | 0.287 (0.025) | 0.391 (0.026)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Stepwise testing of the null hypothesis was used to test the efficacy of Tio R5 and then Tio R2.5, each over placebo. The analysis was performed in a stepwise manner, firstly for this endpoint, then Trough FEV1. Each step was only considered confirmatory if all previous steps were successful; Test type: Superiority or Other; p = 0.2724, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.035, 95% CI 2-sided [-0.028 to 0.099], Standard Error of Mean 0.032 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.139, 95% CI 2-sided [0.075 to 0.203], Standard Error of Mean 0.033 — Difference calculated as Tio R5 minus placebo

2. Secondary Outcome: Trough FEV1 Change From Baseline
Description: Change from baseline in Trough (pre-dose) Forced expiratory volume in 1 second (FEV1) measured at week 12.
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: FAS, missing data at a visit was imputed by the available data from the patient at that visit. Completely missing data were handled by the statistical model.
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 130 | 135 | 128
Litres | 0.136 (0.027) | 0.154 (0.026) | 0.223 (0.027)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Stepwise testing of the null hypothesis was used to test the efficacy of Tio R5 and then Tio R2.5, each over placebo. The analysis for this endpoint was performed in a stepwise manner after the analysis of the primary endpoint was performed. Each step was only considered confirmatory if all previous steps were successful; Test type: Superiority or Other; p = 0.5898, Mixed Models Analysis; Repeated measures restricted maximum likelihood; Mean Difference (Net) = 0.018, 95% CI 2-sided [-0.048 to 0.085], Standard Error of Mean 0.034 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0117, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.087, 95% CI 2-sided [0.019 to 0.154], Standard Error of Mean 0.034 — Difference calculated as Tio R5 minus placebo

3. Secondary Outcome: FVC Peak(0-3h) Change From Baseline
Description: Change from baseline in Maximum forced vital capacity (FVC) measured within the first 3 hours after administration of trial medication (FVC peak(0-3h)) after 12 weeks of treatment.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 130 | 135 | 128
Litres | 0.244 (0.028) | 0.201 (0.027) | 0.275 (0.028)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.2277, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.043, 95% CI 2-sided [-0.113 to 0.027], Standard Error of Mean 0.036 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.3998, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.030, 95% CI 2-sided [-0.040 to 0.101], Standard Error of Mean 0.036 — Difference calculated as Tio R5 minus placebo

4. Secondary Outcome: Trough FVC Change From Baseline
Description: Change from baseline in Trough (pre-dose) FVC measured at week 12.
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 130 | 135 | 128
Litres | 0.141 (0.029) | 0.094 (0.029) | 0.150 (0.030)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.2030, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.048, 95% CI 2-sided [-0.121 to 0.026], Standard Error of Mean 0.037 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.8194, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.009, 95% CI 2-sided [-0.066 to 0.083], Standard Error of Mean 0.038 — Difference calculated as Tio R5 minus placebo

5. Secondary Outcome: FEV1 AUC (0-3h) Change From Baseline
Description: Change from baseline of area under the curve (AUC) from 0 to 3 hours for FEV1 (FEV1 AUC (0-3h)) after 12 weeks of treatment. The AUC was calculated by using the trapezoidal rule divided by the observation time (3h).
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 10 mins before drug administration and 30 mins, 1 hour (h), 2h, 3h after drug administration at 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 130 | 135 | 128
Litres | 0.175 (0.023) | 0.206 (0.022) | 0.301 (0.023)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.2907, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.031, 95% CI 2-sided [-0.026 to 0.088], Standard Error of Mean 0.029 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.126, 95% CI 2-sided [0.068 to 0.184], Standard Error of Mean 0.030 — Difference calculated as Tio R5 minus placebo

6. Secondary Outcome: FVC AUC (0-3h) Change From Baseline
Description: Change from baseline of area under the curve (AUC) from 0 to 3 hours for FVC (Forced vital capacity) (FVC AUC (0-3h)) after 12 weeks of treatment. The AUC was calculated by using the trapezoidal rule divided by the observation time (3h).
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 10 mins before drug administration and 30 mins, 1 hour (h), 2h, 3h after drug administration at 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 130 | 135 | 128
Litres | 0.145 (0.025) | 0.105 (0.024) | 0.182 (0.025)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.2008, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.041, 95% CI 2-sided [-0.103 to 0.022], Standard Error of Mean 0.032 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.2545, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.037, 95% CI 2-sided [-0.026 to 0.100], Standard Error of Mean 0.032 — Difference calculated as Tio R5 minus placebo

7. Secondary Outcome: FEV1 Change From Baseline at Each Individual Timepoint
Description: Forced expiratory volume in one second (FEV1) change from baseline at each individual timepoint.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and 10 mins before drug administration and 30 mins, 1 hour (h), 2h, 3h after drug administration at 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 130 | 135 | 128
Litres
  10 minutes pre-dose | 0.136 (0.027) | 0.154 (0.026) | 0.223 (0.027)
  30 minutes post-dose | 0.166 (0.024) | 0.202 (0.023) | 0.285 (0.024)
  1 hour post-dose | 0.177 (0.025) | 0.203 (0.024) | 0.300 (0.025)
  2 hours post-dose | 0.191 (0.025) | 0.216 (0.025) | 0.324 (0.026)
  3 hours post-dose | 0.168 (0.026) | 0.215 (0.026) | 0.308 (0.026)

8. Secondary Outcome: FVC Change From Baseline at Each Individual Timepoint
Description: FVC change from baseline at each individual timepoint.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and 10 mins before drug administration and 30 mins, 1 hour (h), 2h, 3h after drug administration at 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 130 | 135 | 128
Litres
  10 minutes pre-dose | 0.141 (0.029) | 0.094 (0.029) | 0.150 (0.030)
  30 minutes post-dose | 0.130 (0.026) | 0.096 (0.026) | 0.164 (0.027)
  1 hour post-dose | 0.146 (0.027) | 0.097 (0.026) | 0.181 (0.027)
  2 hours post-dose | 0.159 (0.028) | 0.113 (0.027) | 0.199 (0.028)
  3 hours post-dose | 0.132 (0.028) | 0.110 (0.028) | 0.176 (0.029)

9. Secondary Outcome: Control of Asthma as Assessed by ACQ-IA Total Score
Description: Change from baseline in Interviewer-Administered Asthma Control Questionnaire (ACQ-IA) total score measured at week 12.
  The ACQ-IA is a scale containing 7 questions. Each question has a 7 point scale which ranges from 0 to 6. A score of 0 corresponds to no impairment and a score of 6 corresponds to maximum impairment. ACQ-IA total score is calculated as the mean of the responses to all 7 questions.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 130 | 136 | 126
Units on a scale | 1.026 (0.060) | 1.046 (0.059) | 0.948 (0.061)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.7980, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.020, 95% CI 2-sided [-0.133 to 0.173], Standard Error of Mean 0.078 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.3166, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.079, 95% CI 2-sided [-0.233 to 0.076], Standard Error of Mean 0.079 — Difference calculated as Tio R5 minus placebo

10. Secondary Outcome: ACQ-IA Total Score Responders
Description: Responder categories based on the ACQ-IA total score after 12 weeks of treatment. Analysis was performed using the following categories and definitions: responder (change from trial baseline ≤-0.5), no change (-0.5 <change from trial baseline <0.5) and worsening (change from trial baseline ≥0.5) No statistical testing was performed for ACQ-IA total score responders.
  The ACQ-IA is a scale containing 7 questions, each question has a 7-point scale which ranges from 0 to 6; a score of 0 corresponds to no impairment and a score of 6 corresponds to maximum impairment.
Time Frame: 12 weeks
Population: FAS, missing data for patients not withdrawn from the study were either categorised as no change or based on available data, withdrawn patients were imputed based upon discontinuation reason.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 134 | 136 | 130
Percentage of participants
  Responder | 76.9 | 79.4 | 80.8
  No change | 20.9 | 18.4 | 16.2
  Worsening | 2.2 | 2.2 | 3.1

11. Secondary Outcome: Use of PRN Rescue Medication Per Day
Description: Change from baseline in the number of puffs of rescue medication (salbutamol/albuterol) used per day (24 hour period) based on the weekly mean at week 12.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Number of puffs of rescue medication
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 128 | 136 | 127
Number of puffs of rescue medication | -0.570 (0.096) | -0.553 (0.094) | -0.660 (0.097)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.8916, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.017, 95% CI 2-sided [-0.227 to 0.261], Standard Error of Mean 0.124 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.4789, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.089, 95% CI 2-sided [-0.336 to 0.158], Standard Error of Mean 0.126 — Difference calculated as Tio R5 minus placebo

12. Secondary Outcome: Use of PRN Rescue Medication During the Daytime
Description: Change from baseline in the number of puffs of rescue medication (salbutamol/albuterol) used during the daytime based on the weekly mean at week 12.
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Number of puffs of rescue medication
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 127 | 136 | 126
Number of puffs of rescue medication | -0.279 (0.057) | -0.294 (0.055) | -0.365 (0.057)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.8361, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.015, 95% CI 2-sided [-0.160 to 0.129], Standard Error of Mean 0.074 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.2461, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.087, 95% CI 2-sided [-0.233 to 0.060], Standard Error of Mean 0.075 — Difference calculated as Tio R5 minus placebo

13. Secondary Outcome: Use of PRN Rescue Medication During the Night-time
Description: Change from baseline in the number of puffs of rescue medication (salbutamol/albuterol) used during the night-time based on the weekly mean at week 12.
  Measured values presented are actually adjusted means
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Number of puffs of rescue medication
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 128 | 136 | 126
Number of puffs of rescue medication | -0.285 (0.051) | -0.250 (0.050) | -0.310 (0.052)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.6029, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.035, 95% CI 2-sided [-0.096 to 0.165], Standard Error of Mean 0.067 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.7034, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.026, 95% CI 2-sided [-0.158 to 0.107], Standard Error of Mean 0.067 — Difference calculated as Tio R5 minus placebo

14. Secondary Outcome: Peak Expiratory Flow (PEF) a.m. Change From Baseline
Description: Change from baseline in the morning (a.m.) peak expiratory flow based on the weekly mean at week 12.
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 128 | 136 | 126
L/min | 8.343 (3.613) | 13.119 (3.500) | 13.086 (3.630)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.3083, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 4.776, 95% CI 2-sided [-4.419 to 13.970], Standard Error of Mean 4.686 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.3179, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 4.743, 95% CI 2-sided [-4.571 to 14.057], Standard Error of Mean 4.747 — Difference calculated as Tio R5 minus placebo

15. Secondary Outcome: Peak Expiratory Flow (PEF) p.m. Change From Baseline
Description: Change from baseline in the evening (p.m.) peak expiratory flow based on the weekly mean at week 12.
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 127 | 136 | 126
L/min | 7.892 (3.717) | 8.459 (3.599) | 3.785 (3.731)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.9061, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.567, 95% CI 2-sided [-8.866 to 10.001], Standard Error of Mean 4.807 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.3990, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -4.107, 95% CI 2-sided [-13.658 to 5.444], Standard Error of Mean 4.867 — Difference calculated as Tio R5 minus placebo

16. Secondary Outcome: Peak Expiratory Flow (PEF) Variability Change From Baseline
Description: Change from baseline in the peak expiratory flow variability based on the weekly mean at week 12.
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Percentage of PEF
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 127 | 136 | 125
Percentage of PEF | 0.150 (0.777) | -0.800 (0.749) | -0.352 (0.780)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.3542, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.950, 95% CI 2-sided [-2.959 to 1.060], Standard Error of Mean 1.025 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.6298, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.502, 95% CI 2-sided [-2.545 to 1.541], Standard Error of Mean 1.042 — Difference calculated as Tio R5 minus placebo

17. Secondary Outcome: FEV1 a.m. Change From Baseline
Description: Change from baseline in morning (a.m.) FEV1 based on the weekly mean at week 12.
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 128 | 136 | 126
Litres | 0.174 (0.030) | 0.142 (0.029) | 0.125 (0.030)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.4066, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.032, 95% CI 2-sided [-0.107 to 0.043], Standard Error of Mean 0.038 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.2032, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.049, 95% CI 2-sided [-0.125 to 0.027], Standard Error of Mean 0.039 — Difference calculated as Tio R5 minus placebo

18. Secondary Outcome: FEV1 p.m. Change From Baseline
Description: Change from baseline in evening (p.m.) FEV1 based on the weekly mean at week 12.
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 127 | 136 | 126
Litres | 0.155 (0.031) | 0.104 (0.030) | 0.094 (0.032)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.2064, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.051, 95% CI 2-sided [-0.131 to 0.028], Standard Error of Mean 0.041 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.1410, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.061, 95% CI 2-sided [-0.142 to 0.020], Standard Error of Mean 0.041 — Difference calculated as Tio R5 minus placebo

19. Secondary Outcome: Change From Baseline in Nighttime Awakenings
Description: Change from baseline in nighttime awakenings based on the weekly mean at week 12.
  Nighttime awakenings was assessed by the question "Did you wake up during the night due to your asthma?" from the e-diary. Scores range from 1 (did not wake up) to 5 (was awake all night).
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 128 | 136 | 126
Units on a scale | -0.165 (0.032) | -0.166 (0.031) | -0.159 (0.033)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.9869, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.001, 95% CI 2-sided [-0.083 to 0.082], Standard Error of Mean 0.042 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.8730, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.007, 95% CI 2-sided [-0.077 to 0.090], Standard Error of Mean 0.043 — Difference calculated as Tio R5 minus placebo

20. Secondary Outcome: Change From Baseline in Morning Asthma Symptoms
Description: Change from baseline in morning asthma symptoms based on the weekly mean at week 12.
  Morning asthma symptoms was assessed by the question "how were your asthma symptoms this morning?" from the e-diary. Scores range from 1 (no asthma symptoms) to 5 (very severe asthma symptoms).
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 128 | 136 | 126
Units on a scale | -0.207 (0.038) | -0.213 (0.037) | -0.221 (0.038)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.9043, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.006, 95% CI 2-sided [-0.103 to 0.091], Standard Error of Mean 0.049 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.7708, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.015, 95% CI 2-sided [-0.112 to 0.083], Standard Error of Mean 0.050 — Difference calculated as Tio R5 minus placebo

21. Secondary Outcome: Change From Baseline in Daytime Asthma Symptoms
Description: Change from baseline in daytime asthma symptoms based on the weekly mean at week 12.
  Daytime asthma symptoms was assessed by the question "how were your asthma symptoms during the day?" from the e-diary. Scores range from 1 (no asthma symptoms) to 5 (very severe asthma symptoms).
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 127 | 136 | 126
Units on a scale | -0.226 (0.040) | -0.262 (0.039) | -0.239 (0.041)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.4864, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.036, 95% CI 2-sided [-0.139 to 0.066], Standard Error of Mean 0.052 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.7991, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.013, 95% CI 2-sided [-0.117 to 0.090], Standard Error of Mean 0.053 — Difference calculated as Tio R5 minus placebo

22. Secondary Outcome: Change From Baseline in Daytime Activity Limitations
Description: Change from baseline in daytime activity limitations based on the weekly mean at week 12.
  Daytime activity limitations was assessed by the question "how limited were you in your activities today because of your asthma?" from the e-diary. Scores range from 1 (not limited) to 5 (totally limited).
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 127 | 136 | 126
Units on a scale | -0.210 (0.039) | -0.203 (0.038) | -0.222 (0.039)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.8884, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.007, 95% CI 2-sided [-0.092 to 0.106], Standard Error of Mean 0.050 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.8115, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.012, 95% CI 2-sided [-0.112 to 0.088], Standard Error of Mean 0.051 — Difference calculated as Tio R5 minus placebo

23. Secondary Outcome: Change From Baseline in Daytime Experiences of Shortness of Breath
Description: Change from baseline in daytime experiences of shortness of breath based on the weekly mean at week 12.
  Daytime experiences of shortness of breath was assessed by the question "how much shortness of breath did you experience during the day" from the e-diary. Scores range from 1 (none) to 5 (a very great deal).
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 127 | 136 | 126
Units on a scale | -0.204 (0.039) | -0.187 (0.038) | -0.287 (0.040)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.7498, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.016, 95% CI 2-sided [-0.084 to 0.117], Standard Error of Mean 0.051 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.1108, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.083, 95% CI 2-sided [-0.185 to 0.019], Standard Error of Mean 0.052 — Difference calculated as Tio R5 minus placebo

24. Secondary Outcome: Change From Baseline in Daytime Experiences of Wheeze or Cough
Description: Change from baseline in daytime experiences of wheeze or cough based on the weekly mean at week 12.
  Daytime experiences of wheeze or cough was assessed by the question "did you experience wheeze or cough during the day?" from the e-diary. Scores range from 1 (not at all) to 5 (all the time).
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 127 | 136 | 126
Units on a scale | -0.249 (0.045) | -0.263 (0.044) | -0.320 (0.046)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.8055, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.015, 95% CI 2-sided [-0.131 to 0.102], Standard Error of Mean 0.059 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.2360, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.071, 95% CI 2-sided [-0.189 to 0.047], Standard Error of Mean 0.060 — Difference calculated as Tio R5 minus placebo

25. Secondary Outcome: Change From Baseline in Asthma Symptom-free Days
Description: Change from baseline in asthma symptom-free days based on the weekly mean at week 12.
  A day was considered as an asthma symptom-free day if there were no symptoms reported via the e-Diary and no use of rescue medication reported via the eDiary during that day.
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 128 | 136 | 127
Days | 0.147 (0.031) | 0.130 (0.030) | 0.172 (0.031)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.6748, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.017, 95% CI 2-sided [-0.097 to 0.063], Standard Error of Mean 0.041 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.5497, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.025, 95% CI 2-sided [-0.056 to 0.105], Standard Error of Mean 0.041 — Difference calculated as Tio R5 minus placebo

ADVERSE EVENTS:
Time Frame: From first drug intake until 30 days after last drug intake, up to 164 days
Description: The final study visit was postponed if the status of the patient could affect the primary endpoint, for example, in cases of asthma exacerbations, therefore patients could remain on treatment for longer than the planned 12 weeks.
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Serious Adverse Events (participants affected / at risk) | 2/134 | 2/136 | 4/130
Other Adverse Events (participants affected / at risk) | 49/134 | 36/136 | 35/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Respimat (N=134) | Tio R2.5 (N=136) | Tio R5 (N=130)
Appendicitis (Infections and infestations) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Respimat (N=134) | Tio R2.5 (N=136) | Tio R5 (N=130)
Nasopharyngitis (Infections and infestations) | 11 | 6 | 6
Peak expiratory flow rate decreased (Investigations) | 20 | 15 | 15
Asthma (Respiratory, thoracic and mediastinal disorders) | 29 | 20 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.